CLINICAL TRIAL: NCT01666496
Title: An Interactive Video Game for HIV Prevention in Early Adolescents
Brief Title: An Interactive Game for HIV Prevention in Early Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Principal Investigator, Lynn E. Fiellin, Associate Professor, Yale University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1208010715
Record Dates: First submitted 2012-08-09; First posted 2012-08-16 (Estimated); Last update posted 2017-06-27 (Actual); Status verified 2017-02

CONDITIONS: HIV; Risk Reduction
Keywords: Adolescent; risk; HIV; video games
MeSH Terms: conditions — Risk Reduction Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental Video Game (Experimental): Participants will play the experimental videogame for 6 weeks. The intervention will be provided during 12 sessions, twice weekly for 6 weeks; each session will involve one and one-quarter hour of game play.
  Interventions: Behavioral: Experimental Video Game
- Off the Shelf Video Game (Other): Participants will play the off the shelf videogame for 6 weeks. The intervention be provided during 12 sessions, twice weekly for 6 weeks; each session will involve one and one-quarter hour of game play.
  Interventions: Behavioral: Off the Shelf Video Game

INTERVENTIONS:
Behavioral: Experimental Video Game — Participants will play either the experimental or the control videogame for 6 weeks. Both interventions will be provided during 12 sessions, twice weekly for 6 weeks; each session will involve one and one-quarter hour of game play.
  Arms: Experimental Video Game
Behavioral: Off the Shelf Video Game — Participants will play either the experimental or the control videogame for 6 weeks. Both interventions will be provided during 12 sessions, twice weekly for 6 weeks; each session will involve one and one-quarter hour of game play.
  Arms: Off the Shelf Video Game

SUMMARY:
The purpose of this study is to evaluate, through a randomized clinical trial, the efficacy of an interactive video game the investigators are developing at reducing risk behaviors in at-risk teens.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate, through a randomized clinical trial, the efficacy of an interactive video game the investigators are developing at reducing risk behaviors in at-risk teens. The investigators are using proven components of HIV prevention interventions, social cognitive theory, self-efficacy, prospect theory, message framing, and video gaming principles to develop and evaluate this interactive HIV prevention video game. In Phase 1 of this project, the investigators have been working with Schell Games of Pittsburgh, PA, Digitalmill of Portland, ME, and the Farnam Neighborhood House in New Haven, CT to develop our interactive video game with the input from our experts and focus groups and interviews with adolescents. Phase 1 has been a developmental iterative process in which the investigators have been building the software for the game for the purposes of targeting HIV prevention in our population of interest: young minority adolescents. Following development of the video game, the investigators will move to Phase 2 in which the investigators will enroll 330 minority adolescents who are attendees at one of several after-school programs in the greater New Haven area and assign them to play either the experimental game or a control game. In the experimental game, the player will be presented with a series of "risk challenges" thereby helping them to develop sex, drug and alcohol negotiation and refusal skills.

ELIGIBILITY:
Inclusion Criteria:

1. Ages 11-14 years
2. Able to provide assent/parental/guardian consent
3. Agree to participate in a computer-based videogame (willing to sit at a computer for 75 minutes twice weekly to play the game)
4. English-speaking

Exclusion Criteria:

1. Not between the ages of 11-14 years
2. Not able to provide assent/parental/guardian consent
3. Not willing to sit at a computer for 75 minutes twice weekly to play the game
4. Non-English speaking

Ages: 11 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 333 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2016-06-18 (Actual); Study Completion 2016-06-18 (Actual)

PRIMARY OUTCOMES:
Delay in the initiation of sexual activity | 3 weeks
  The primary outcome measure will be delay in initiating sexual activity. Delay in initiation of sexual activity will be defined as individuals who report having never had voluntary sexual intercourse prior to the baseline assessment and continue to not initiate sexual activity. Those who report initiating sex between baseline and the follow-up period are defined as having initiated sexual activity.
Delay in the initiation of sexual activity | 6 weeks
  The primary outcome measure will be delay in initiating sexual activity. Delay in initiation of sexual activity will be defined as individuals who report having never had voluntary sexual intercourse prior to the baseline assessment and continue to not initiate sexual activity. Those who report initiating sex between baseline and the follow-up period are defined as having initiated sexual activity.
Delay in the initiation of sexual activity | 3 months
  The primary outcome measure will be delay in initiating sexual activity. Delay in initiation of sexual activity will be defined as individuals who report having never had voluntary sexual intercourse prior to the baseline assessment and continue to not initiate sexual activity. Those who report initiating sex between baseline and the follow-up period are defined as having initiated sexual activity.
Delay in the initiation of sexual activity | 6 months
  The primary outcome measure will be delay in initiating sexual activity. Delay in initiation of sexual activity will be defined as individuals who report having never had voluntary sexual intercourse prior to the baseline assessment and continue to not initiate sexual activity. Those who report initiating sex between baseline and the follow-up period are defined as having initiated sexual activity.
Delay in the initiation of sexual activity | 12 months
  The primary outcome measure will be delay in initiating sexual activity. Delay in initiation of sexual activity will be defined as individuals who report having never had voluntary sexual intercourse prior to the baseline assessment and continue to not initiate sexual activity. Those who report initiating sex between baseline and the follow-up period are defined as having initiated sexual activity.
Delay in the initiation of sexual activity | 24 months
  The primary outcome measure will be delay in initiating sexual activity. Delay in initiation of sexual activity will be defined as individuals who report having never had voluntary sexual intercourse prior to the baseline assessment and continue to not initiate sexual activity. Those who report initiating sex between baseline and the follow-up period are defined as having initiated sexual activity.

SECONDARY OUTCOMES:
Knowledge about HIV/AIDS risk behaviors and transmission | 3 weeks
  To determine if an interactive videogame focused on developing sex, drug and alcohol negotiation and refusal skills, compared to a control game, increases HIV risk knowledge in minority early adolescents.
Level of social competency in using negotiating and refusal skills in the virtual environment | 3 weeks
  To determine if an interactive videogame focused on developing sex, drug and alcohol negotiation and refusal skills, compared to a control game, increases social competency in using negotiating and refusal skills in the virtual environment in minority early adolescents. Social competency is defined as skills that allow the individual to achieve personal goals in social interaction while maintaining positive relationships with others over time and across situations. This will be captured through data collected during the game play, including the participant's ability to negotiate social situations and successfully refuse risky situations.
Level of self-efficacy regarding negotiation around initiation of sexual activity | 3 weeks
  To determine if an interactive videogame focused on developing sex, drug and alcohol negotiation and refusal skills, compared to a control game, increases self-efficacy regarding negotiation around initiation of sexual activity in minority adolescents.We will use 7 items to assess self-efficacy to refuse sexual behaviors. Participants will be presented with the situation "imagine you are alone with someone you like very much" and then asked to indicate how confident they are that they could stop the person if he or she wanted to (a) kiss them on the lips, (b) touch their chest or breasts, (c) touch their private parts below the waist, (d) have oral sex, or (e) have vaginal sex. Participants will report how confident they are that they could refuse sex if they had been drinking or had strong sexual feelings for someone. Self-efficacy for condom use will be measured using 5 items (e.g., "If you wanted to get a condom, how sure are you that you could go to the store and buy one?").
Drug and alcohol use behaviors | 3 weeks
  To determine if an interactive videogame focused on developing sex, drug and alcohol negotiation and refusal skills, compared to a control game, decreases drug and alcohol use behaviors in minority early adolescents.
Level of self-efficacy in negotiating situations involving offers of drugs and alcohol | 3 weeks
  To determine if an interactive videogame focused on developing sex, drug and alcohol negotiation and refusal skills, compared to a control game, increases self-efficacy in negotiating situations involving offers of drugs and alcohol in minority adolescents.To assess participants' self-efficacy to refuse drugs we will use 6 items adapted from the Drug Use Resistance Self-Efficacy (DURSE) Scale for Young Adolescents (Carpenter & Howard, 2009). We will administer 2 items each for cigarettes, alcohol, and marijuana assessing participants' confidence to refuse the drug if it is offered by (a) a friend or (b) an older friend of family member.
Overall risk-taking behaviors | 3 weeks
  To determine if an interactive videogame focused on developing sex, drug and alcohol negotiation and refusal skills, compared to a control game,reduces overall risk-taking behaviors in minority early adolescents.
Knowledge about HIV/AIDS risk behaviors and transmission | 6 weeks
  To determine if an interactive videogame focused on developing sex, drug and alcohol negotiation and refusal skills, compared to a control game, increases HIV risk knowledge in minority early adolescents.
Knowledge about HIV/AIDS risk behaviors and transmission | 3 months
  To determine if an interactive videogame focused on developing sex, drug and alcohol negotiation and refusal skills, compared to a control game, increases HIV risk knowledge in minority early adolescents.
Knowledge about HIV/AIDS risk behaviors and transmission | 6 months
  To determine if an interactive videogame focused on developing sex, drug and alcohol negotiation and refusal skills, compared to a control game, increases HIV risk knowledge in minority early adolescents.
Knowledge about HIV/AIDS risk behaviors and transmission | 12 months
  To determine if an interactive videogame focused on developing sex, drug and alcohol negotiation and refusal skills, compared to a control game, increases HIV risk knowledge in minority early adolescents.
Knowledge about HIV/AIDS risk behaviors and transmission | 24 months
  To determine if an interactive videogame focused on developing sex, drug and alcohol negotiation and refusal skills, compared to a control game, increases HIV risk knowledge in minority early adolescents.
Level of social competency in using negotiating and refusal skills in the virtual environment | 6 weeks
  To determine if an interactive videogame focused on developing sex, drug and alcohol negotiation and refusal skills, compared to a control game, increases social competency in using negotiating and refusal skills in the virtual environment in minority early adolescents.Social competency is defined as skills that allow the individual to achieve personal goals in social interaction while maintaining positive relationships with others over time and across situations. This will be captured through data collected during the game play, including the participant's ability to negotiate social situations and successfully refuse risky situations.
Level of social competency in using negotiating and refusal skills in the virtual environment | 3 months
  To determine if an interactive videogame focused on developing sex, drug and alcohol negotiation and refusal skills, compared to a control game, increases social competency in using negotiating and refusal skills in the virtual environment in minority early adolescents.Social competency is defined as skills that allow the individual to achieve personal goals in social interaction while maintaining positive relationships with others over time and across situations. This will be captured through data collected during the game play, including the participant's ability to negotiate social situations and successfully refuse risky situations.
Level of social competency in using negotiating and refusal skills in the virtual environment | 6 months
  To determine if an interactive videogame focused on developing sex, drug and alcohol negotiation and refusal skills, compared to a control game, increases social competency in using negotiating and refusal skills in the virtual environment in minority early adolescents.Social competency is defined as skills that allow the individual to achieve personal goals in social interaction while maintaining positive relationships with others over time and across situations. This will be captured through data collected during the game play, including the participant's ability to negotiate social situations and successfully refuse risky situations.
Level of social competency in using negotiating and refusal skills in the virtual environment | 12 months
  To determine if an interactive videogame focused on developing sex, drug and alcohol negotiation and refusal skills, compared to a control game, increases social competency in using negotiating and refusal skills in the virtual environment in minority early adolescents. Social competency is defined as skills that allow the individual to achieve personal goals in social interaction while maintaining positive relationships with others over time and across situations. This will be captured through data collected during the game play, including the participant's ability to negotiate social situations and successfully refuse risky situations.
Level of social competency in using negotiating and refusal skills in the virtual environment | 24 months
  To determine if an interactive videogame focused on developing sex, drug and alcohol negotiation and refusal skills, compared to a control game, increases social competency in using negotiating and refusal skills in the virtual environment in minority early adolescents.Social competency is defined as skills that allow the individual to achieve personal goals in social interaction while maintaining positive relationships with others over time and across situations. This will be captured through data collected during the game play, including the participant's ability to negotiate social situations and successfully refuse risky situations.
Level of self-efficacy regarding negotiation around initiation of sexual activity | 6 weeks
  To determine if an interactive videogame focused on developing sex, drug and alcohol negotiation and refusal skills, compared to a control game, increases self-efficacy regarding negotiation around initiation of sexual activity in minority adolescents.We will use 7 items to assess self-efficacy to refuse sexual behaviors. Participants will be presented with the situation "imagine you are alone with someone you like very much" and then asked to indicate how confident they are that they could stop the person if he or she wanted to (a) kiss them on the lips, (b) touch their chest or breasts, (c) touch their private parts below the waist, (d) have oral sex, or (e) have vaginal sex. Participants will report how confident they are that they could refuse sex if they had been drinking or had strong sexual feelings for someone. Self-efficacy for condom use will be measured using 5 items (e.g., "If you wanted to get a condom, how sure are you that you could go to the store and buy one?").
Level of self-efficacy regarding negotiation around initiation of sexual activity | 3 months
  To determine if an interactive videogame focused on developing sex, drug and alcohol negotiation and refusal skills, compared to a control game, increases self-efficacy regarding negotiation around initiation of sexual activity in minority adolescents.We will use 7 items to assess self-efficacy to refuse sexual behaviors. Participants will be presented with the situation "imagine you are alone with someone you like very much" and then asked to indicate how confident they are that they could stop the person if he or she wanted to (a) kiss them on the lips, (b) touch their chest or breasts, (c) touch their private parts below the waist, (d) have oral sex, or (e) have vaginal sex. Participants will report how confident they are that they could refuse sex if they had been drinking or had strong sexual feelings for someone. Self-efficacy for condom use will be measured using 5 items (e.g., "If you wanted to get a condom, how sure are you that you could go to the store and buy one?").
Level of self-efficacy regarding negotiation around initiation of sexual activity | 6 months
  To determine if an interactive videogame focused on developing sex, drug and alcohol negotiation and refusal skills, compared to a control game, increases self-efficacy regarding negotiation around initiation of sexual activity in minority adolescents.We will use 7 items to assess self-efficacy to refuse sexual behaviors. Participants will be presented with the situation "imagine you are alone with someone you like very much" and then asked to indicate how confident they are that they could stop the person if he or she wanted to (a) kiss them on the lips, (b) touch their chest or breasts, (c) touch their private parts below the waist, (d) have oral sex, or (e) have vaginal sex. Participants will report how confident they are that they could refuse sex if they had been drinking or had strong sexual feelings for someone. Self-efficacy for condom use will be measured using 5 items (e.g., "If you wanted to get a condom, how sure are you that you could go to the store and buy one?").
Level of self-efficacy regarding negotiation around initiation of sexual activity | 12 months
  To determine if an interactive videogame focused on developing sex, drug and alcohol negotiation and refusal skills, compared to a control game, increases self-efficacy regarding negotiation around initiation of sexual activity in minority adolescents.We will use 7 items to assess self-efficacy to refuse sexual behaviors. Participants will be presented with the situation "imagine you are alone with someone you like very much" and then asked to indicate how confident they are that they could stop the person if he or she wanted to (a) kiss them on the lips, (b) touch their chest or breasts, (c) touch their private parts below the waist, (d) have oral sex, or (e) have vaginal sex. Participants will report how confident they are that they could refuse sex if they had been drinking or had strong sexual feelings for someone. Self-efficacy for condom use will be measured using 5 items (e.g., "If you wanted to get a condom, how sure are you that you could go to the store and buy one?").
Level of self-efficacy regarding negotiation around initiation of sexual activity | 24 months
  To determine if an interactive videogame focused on developing sex, drug and alcohol negotiation and refusal skills, compared to a control game, increases self-efficacy regarding negotiation around initiation of sexual activity in minority adolescents.We will use 7 items to assess self-efficacy to refuse sexual behaviors. Participants will be presented with the situation "imagine you are alone with someone you like very much" and then asked to indicate how confident they are that they could stop the person if he or she wanted to (a) kiss them on the lips, (b) touch their chest or breasts, (c) touch their private parts below the waist, (d) have oral sex, or (e) have vaginal sex. Participants will report how confident they are that they could refuse sex if they had been drinking or had strong sexual feelings for someone. Self-efficacy for condom use will be measured using 5 items (e.g., "If you wanted to get a condom, how sure are you that you could go to the store and buy one?").
Drug and alcohol use behaviors | 6 weeks
  To determine if an interactive videogame focused on developing sex, drug and alcohol negotiation and refusal skills, compared to a control game, decreases drug and alcohol use behaviors in minority early adolescents.
Drug and alcohol use behaviors | 3 months
  To determine if an interactive videogame focused on developing sex, drug and alcohol negotiation and refusal skills, compared to a control game, decreases drug and alcohol use behaviors in minority early adolescents.
Drug and alcohol use behaviors | 6 months
  To determine if an interactive videogame focused on developing sex, drug and alcohol negotiation and refusal skills, compared to a control game, decreases drug and alcohol use behaviors in minority early adolescents.
Drug and alcohol use behaviors | 12 months
  To determine if an interactive videogame focused on developing sex, drug and alcohol negotiation and refusal skills, compared to a control game, decreases drug and alcohol use behaviors in minority early adolescents.
Drug and alcohol use behaviors | 24 months
  To determine if an interactive videogame focused on developing sex, drug and alcohol negotiation and refusal skills, compared to a control game, decreases drug and alcohol use behaviors in minority early adolescents.
Level of self-efficacy in negotiating situations involving offers of drugs and alcohol | 6 weeks
  To determine if an interactive videogame focused on developing sex, drug and alcohol negotiation and refusal skills, compared to a control game, increases self-efficacy in negotiating situations involving offers of drugs and alcohol in minority adolescents.To assess participants' self-efficacy to refuse drugs we will use 6 items adapted from the Drug Use Resistance Self-Efficacy (DURSE) Scale for Young Adolescents (Carpenter & Howard, 2009). We will administer 2 items each for cigarettes, alcohol, and marijuana assessing participants' confidence to refuse the drug if it is offered by (a) a friend or (b) an older friend of family member.
Level of self-efficacy in negotiating situations involving offers of drugs and alcohol | 3 months
  To determine if an interactive videogame focused on developing sex, drug and alcohol negotiation and refusal skills, compared to a control game, increases self-efficacy in negotiating situations involving offers of drugs and alcohol in minority adolescents.To assess participants' self-efficacy to refuse drugs we will use 6 items adapted from the Drug Use Resistance Self-Efficacy (DURSE) Scale for Young Adolescents (Carpenter & Howard, 2009). We will administer 2 items each for cigarettes, alcohol, and marijuana assessing participants' confidence to refuse the drug if it is offered by (a) a friend or (b) an older friend of family member.
Level of self-efficacy in negotiating situations involving offers of drugs and alcohol | 6 months
  To determine if an interactive videogame focused on developing sex, drug and alcohol negotiation and refusal skills, compared to a control game, increases self-efficacy in negotiating situations involving offers of drugs and alcohol in minority adolescents.To assess participants' self-efficacy to refuse drugs we will use 6 items adapted from the Drug Use Resistance Self-Efficacy (DURSE) Scale for Young Adolescents (Carpenter & Howard, 2009). We will administer 2 items each for cigarettes, alcohol, and marijuana assessing participants' confidence to refuse the drug if it is offered by (a) a friend or (b) an older friend of family member.
Level of self-efficacy in negotiating situations involving offers of drugs and alcohol | 12 months
  To determine if an interactive videogame focused on developing sex, drug and alcohol negotiation and refusal skills, compared to a control game, increases self-efficacy in negotiating situations involving offers of drugs and alcohol in minority adolescents.To assess participants' self-efficacy to refuse drugs we will use 6 items adapted from the Drug Use Resistance Self-Efficacy (DURSE) Scale for Young Adolescents (Carpenter & Howard, 2009). We will administer 2 items each for cigarettes, alcohol, and marijuana assessing participants' confidence to refuse the drug if it is offered by (a) a friend or (b) an older friend of family member.
Level of self-efficacy in negotiating situations involving offers of drugs and alcohol | 24 months
  To determine if an interactive videogame focused on developing sex, drug and alcohol negotiation and refusal skills, compared to a control game, increases self-efficacy in negotiating situations involving offers of drugs and alcohol in minority adolescents.To assess participants' self-efficacy to refuse drugs we will use 6 items adapted from the Drug Use Resistance Self-Efficacy (DURSE) Scale for Young Adolescents (Carpenter & Howard, 2009). We will administer 2 items each for cigarettes, alcohol, and marijuana assessing participants' confidence to refuse the drug if it is offered by (a) a friend or (b) an older friend of family member.
Overall risk-taking behaviors | 6 weeks
  To determine if an interactive videogame focused on developing sex, drug and alcohol negotiation and refusal skills, compared to a control game,reduces overall risk-taking behaviors in minority early adolescents.
Overall risk-taking behaviors | 3 months
  To determine if an interactive videogame focused on developing sex, drug and alcohol negotiation and refusal skills, compared to a control game,reduces overall risk-taking behaviors in minority early adolescents.
Overall risk-taking behaviors | 6 months
  To determine if an interactive videogame focused on developing sex, drug and alcohol negotiation and refusal skills, compared to a control game,reduces overall risk-taking behaviors in minority early adolescents.
Overall risk-taking behaviors | 12 months
  To determine if an interactive videogame focused on developing sex, drug and alcohol negotiation and refusal skills, compared to a control game,reduces overall risk-taking behaviors in minority early adolescents.
Overall risk-taking behaviors | 24 months
  To determine if an interactive videogame focused on developing sex, drug and alcohol negotiation and refusal skills, compared to a control game,reduces overall risk-taking behaviors in minority early adolescents.

CONTACTS AND LOCATIONS:
Overall Officials: Lynn E Fiellin, MD, Principal Investigator — Yale University
Locations (1):
- Yale School of Medicine, New Haven, Connecticut, United States

REFERENCES:
- [Derived] Fiellin LE, Hieftje KD, Pendergrass TM, Kyriakides TC, Duncan LR, Dziura JD, Sawyer BG, Mayes L, Crusto CA, Forsyth BW, Fiellin DA. Video Game Intervention for Sexual Risk Reduction in Minority Adolescents: Randomized Controlled Trial. J Med Internet Res. 2017 Sep 18;19(9):e314. doi: 10.2196/jmir.8148. PMID 28923788
- [Derived] Montanaro E, Fiellin LE, Fakhouri T, Kyriakides TC, Duncan LR. Using Videogame Apps to Assess Gains in Adolescents' Substance Use Knowledge: New Opportunities for Evaluating Intervention Exposure and Content Mastery. J Med Internet Res. 2015 Oct 28;17(10):e245. doi: 10.2196/jmir.4377. PMID 26510775
- See also: Related info — http://www.play2prevent.org